CLINICAL TRIAL: NCT03646799
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability After Oral Administration of CKD-387 10/1000 mg and D484 10/1000mg in Healthy Adults
Brief Title: Pharmacokinetics and Safety/Tolerability After Oral Administration of CKD-387 and D484 in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 184BE18012
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Period 1: 1 tablet of reference drug(D484) Period 2: 1 tablet of test drug(CKD-387)
  Interventions: Drug: CKD-387; Drug: D484
- Group 2 (Experimental): Period 1: 1 tablet of test drug(CKD-387) Period 2: 1 tablet of reference drug(D484)
  Interventions: Drug: CKD-387; Drug: D484

INTERVENTIONS:
Drug: CKD-387 — test drug
Drug: D484 — reference drug

SUMMARY:
Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability after Oral Administration of CKD-387 10/1000 mg and D484 10/1000mg in Healthy Adults

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 19 and 55
* Body weight ≥ 55kg for male, ≥ 50kg for female
* Body mass index ≥ 18.5 kg/m2 and < 25.0 kg/m2
* Females who are post-menopausal or underwent sterilization
* Males who agreed to practice contraception until after 28 days of last intake Investigational product
* Ability to provide written informed consent

Exclusion Criteria:

* Subject with clinically significant hepatic, renal, nervous, immune, respiratory, endocrine, hemato-oncology, cardiovascular systemic disease and psychosis disorder
* Subject who are weak in dehydration or clinically significant dehydration
* IV injecting examination of radioactive-iodine substances within 48 hours prior to first IP administration
* Subjects who have Galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Subjects with history of gastrointestinal disease or surgery that may affect absorption of IP
* Hypersensitive to dapagliflozin/metformin
* At screening,

  * AST(Aspartate Transaminase), ALT(Alanine Transaminase) > UNL(upper normal limit)*1.25
  * Total Bilirubin > UNL(upper normal limit)*1.5, CPK > UNL(upper normal limit)*1.5
  * eGFR(estimated Glomerular Filtration Rate) < 60 mL/min/1.73m2(Modification of diet in renal Disease calculated)
  * Positive reaction on following tests: Hepatitis B, Hepatitis C, HIV(Human Immunodeficiency Virus) and syphilis
  * SBP(Systolic blood pressure) ≥ 150 mmHg or < 90 mmHg, DBP(Diastolic blood pressure) > 100 mmHg or < 50 mmHg
* History of drug abuse or positive urine drug screening results
* Women with pregnant, breast-feeding
* Caffeine > 5 cups/day, Alcohol > 210 g/week, Smoker > 10 cigarettes /day or who are unable to stop caffeine intake, drinking alcohol and smoking until the last blood drawing for PK
* Subject who took ethical drug/herbal compound within 14 days, over-the-counter drug/vitamin supplements within 7 days and depot injection/implantation within 30 days prior to the first IP administration
* Subject who was enrolled in another clinical trial(including Bioequivalence study) and administered drugs within 90 days prior to the first IP administration
* Subject with whole blood donation within 60 days or component blood donation within 30 days
* Not eligible to participate for the study at the discretion of Investigator

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-08-30 (Estimated); Primary Completion 2018-09-09 (Estimated); Study Completion 2018-09-14 (Estimated)

PRIMARY OUTCOMES:
Cmax of Dapagliflozin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Maximum plasma concentration of Dapagliflozin
Cmax of Metformin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Maximum plasma concentration of Metformin
AUClast of Dapagliflozin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Area under the plasma concentration-time curve to last concentration of Dapagliflozin
AUClast of Metformin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Area under the plasma concentration-time curve to last concentration of Metformin

SECONDARY OUTCOMES:
AUCinf of Dapagliflozin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Area under the plasma concentration-time curve from zero to infinity concentration of Dapagliflozin
AUCinf of Metformin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Area under the plasma concentration-time curve from zero to infinity concentration of Metformin
Tmax of Dapagliflozin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Time to maximum plasma concentration of Dapagliflozin
Tmax of Metformin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Time to maximum plasma concentration of Metformin
T1/2 of Dapagliflozin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Half-life of Dapagliflozin
T1/2 of Metformin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Half-life of Metformin
Vd/F of Dapagliflozin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Apparent volume of distribution of Dapagliflozin
Vd/F of Metformin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Apparent volume of distribution of Metformin
CL/F of Dapagliflozin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Apparent clearance of Dapagliflozin
CL/F of Metformin | Predose(0h), 0.33, 0.67, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 32, and 48 hour after drug administration
  Apparent clearance of Metformin

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Severance Hospital, Soeul, South Korea